CLINICAL TRIAL: NCT02945540
Title: Assessment of Patient Satisfaction Supported in the Patient Education Program "Gestational Diabetes" at the University Hospital of Caen
Brief Title: Assessment of Patient Satisfaction Program "Gestational Diabetes"
Acronym: SATISFYDG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-198
Record Dates: First submitted 2016-08-25; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; Patient education; Patient Satisfaction
MeSH Terms: conditions — Diabetes, Gestational; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study seeks to evaluate patient satisfaction within the patient therapeutic education program "gestational diabetes" (multidisciplinary and multi-professional program) to see if they deem effective to limit the impact of gestational diabetes on pregnancy . Patients are questioned on the skills acquired in everyday life, the effective support in personal development, development of self-determination capabilities and communication with health professionals.

This study must include all patients participating in the therapeutic education program for a year and meeting the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* Gestational diabetes diagnosis based on OGTT glucose 75g, performed after 24 weeks of gestation
* Women aged 18 and over
* After 24th week of gestation
* Before 36th week of gestation
* initial management in therapeutic education at the University Hospital of Caen

Exclusion Criteria:

* Another form of diabetes (existing before pregnancy or diagnosed before 24 weeks of gestation)
* women under 18 years
* Initial management of gestational diabetes by health professionals outside the University Hospital of Caen
* Poor understanding of the French language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with gestational diabetes and cared in therapeutic patient education
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Measuring patient satisfaction by a questionnaire on therapeutic education | 36th week of gestation
  Evaluation of satisfaction the entry into the program, after the diagnosis, until the 36th week of gestation.
Measuring patient satisfaction at childbirth by a questionnaire on satisfaction of hospital care | baseline
  Assessment of satisfaction between the 36th week of gestation and childbirth.

SECONDARY OUTCOMES:
Blood glucose self-monitoring | until birth (up to a maximum of 16 weeks)
  control of diabetes by expected blood glucose targets
weight gain | during pregnancy until birth (up to a maximum of 16 weeks)
type of birth | baseline
  Mode of parturition : Cesarean section or vaginal birth
Measure of abdominal diameter | before childbirth
  Fetal Macrosomia suspected during fetal ultrasonography
Measure of fetal weight | before childbirth
  Fetal Macrosomia suspected during fetal ultrasonography
Birth weight | at childbirth
Apgar score | 1 minute and 5 minutes after birthchild
Neonatal blood glucose measurement | during the first 48 hours after birth
  Number of neonatal hypoglycemia

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No